CLINICAL TRIAL: NCT03257085
Title: CALIBER (Carbohydrates, Lipids and Biomarkers of Traditional and Emerging Cardiometabolic Risk Factors) Phase 1: A Pilot Study in Normal-weight and Overweight Adults.
Brief Title: CALIBER Phase 1: A Pilot Study in Normal-weight and Overweight Adults.
Acronym: CALIBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Hope University (Other)
Responsible Party: Principal Investigator, Tanja Harrison, PhD Researcher and Registered Associate Nutritionist, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CALIBER
Record Dates: First submitted 2017-08-14; First posted 2017-08-22 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Cardiometabolic Risk

STUDY DESIGN:
Intervention Model Description: Randomised pilot study
Masking Description: Due to the nature of the low-carbohydrate, high-fat and high-carbohydrate, moderate-fat diets masking is not feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate, high-fat (Experimental): Participants adhering to low-carbohydrate, high-fat diet for 8 weeks.
  Interventions: Other: Low-carbohydrate, high-fat
- High-carbohydrate, moderate fat (Experimental): Participants following high-carbohydrate, moderate-fat diet for 8 weeks.
  Interventions: Other: High-carbohydrate, moderate-fat

INTERVENTIONS:
Other: Low-carbohydrate, high-fat — Participants following low-carbohydrate, high-fat diet for 8 weeks.
  Other Names: CALIBER LCHF
  Arms: Low-carbohydrate, high-fat
Other: High-carbohydrate, moderate-fat — Participants following high-carbohydrate, moderate-fat diet (UK dietary guidelines) for 8 weeks.
  Other Names: CALIBER HCMF
  Arms: High-carbohydrate, moderate fat

SUMMARY:
Pilot study to compare the impact of following a low-carbohydrate, high-fat diet versus following a high-carbohydrates, moderate-fat diet (UK dietary guidelines) on cardiometabolic risk markers and associated behaviours in a normal-weight and overweight adult population.

DETAILED DESCRIPTION:
Cardiometabolic diseases (CMD), such as type 2 diabetes and cardiovascular disease (CVD), are globally amongst the highest contributors to morbidity and mortality with high (cost) implications to the overall economy and health care systems. A number of risk markers have been associated with CMDs, including blood serum markers, low levels of lean mass and high levels of body fat, including increased waist circumference. Dietary factors and nutritional status have long been linked with specific markers of cardiometabolic (CM) risk. The quantity and quality of dietary carbohydrates has been associated with increased serum triglycerides levels, increased body fat mass, increased waist circumference and visceral fat around the organs in particular. They also seem to increase food cravings. Whilst official dietary guidelines in the UK and elsewhere still recommend a high carbohydrate and low fat diet as standard, these recommendations have increasingly been challenged. Evidence has been mounting that very-low carbohydrate (ketogenic) and low carbohydrate diets can ameliorate CM risk factors, especially when a personalised rather than a one-size-fits-all approach is being taken. Response to carbohydrate load and adherence to dietary interventions can vary widely dependent on individual substrate and energy metabolism and insulin-resistant status.

The majority of dietary interventions with ketogenic and low-carbohydrate diets has focused on weight loss as the primary outcome in overweight and obese individuals. However, in recent years evidence has been mounting that the location and quality of adipose tissue (AT) play a more important role in manifestation of CM risk than quantity of AT alone. Detrimental health behaviours, such as low-quality diet and low levels of physical activity seem to be important contributors to this.

Further studies can provide vital insights into the links between diet, location-specific adipose tissue, CM risk factors and health-related behaviours.

Therefore this 8-weeks randomised pilot study will investigate the impact of either following a low-carbohydrate, high-fat diet versus following a high-carbohydrates, moderate-fat diet (UK dietary guidelines) on cardiometabolic risk markers and associated behaviours in a normal-weight and overweight adult population aged 19 - 64 at potential risk of CMD.

ELIGIBILITY:
Inclusion Criteria cohort 1:

1. BMI 18.5 - 29.9kg/m2
2. Aged 19 - 64
3. White-Caucasian
4. Score of ≥4 from a combination of risk markers, including

   * Fasting glucose concentration >5.5mmol/L = 3 points
   * Waist >102cm or 40 inches = 2 points (males)
   * Waist >94 cm or 37 inches = 1 point (males)
   * Waist >88cm or 34inches = 2 points (females)
   * Waist >80 cm or 31 inches = 1 point (females)
   * Systolic blood pressure>130mmHg = 1 point
   * Diastolic BP >85mmHg = 1 point
   * HDL cholesterol concentration <1.0mmol/L = 2 points
   * Serum triglyceride concentration >1.3mmol/L = 1 point.

Exclusion Criteria cohort 1:

1. Smoker
2. Vegetarian or vegan
3. Suffering from food allergies or intolerances
4. Drinking alcohol above recommended UK government guidelines
5. Previous diagnosis of CM disease
6. Taking lipid-lowering medication
7. Taking blood pressure-lowering medication
8. Taking blood glucose-lowering medication
9. Taking dietary supplements
10. Suffering from an eating disorder
11. Current or previous renal impairment

Inclusion Criteria cohort 2:

1. BMI 18.5 - 29.9kg/m2
2. Aged 19 - 64
3. White-Caucasian

Exclusion Criteria cohort 2:

1. Smoker
2. Vegetarian or vegan
3. Suffering from food allergies or intolerances
4. Drinking alcohol above recommended UK government guidelines
5. Previous diagnosis of CM disease
6. Taking lipid-lowering medication
7. Taking blood pressure-lowering medication
8. Taking blood glucose-lowering medication
9. Taking dietary supplements
10. Suffering from an eating disorder
11. Current or previous renal impairment

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Serum lipid profile | 8 weeks
  Total cholesterol, HDL-C, LDL-C, non-HDL cholesterol, small-dense LDL-C and triglycerides measured in mmol/L
Blood glucose | 8 weeks
  Measured in mmol/L
Systolic and diastolic blood pressure | 8 weeks
  Measured in mmHg
Inflammatory markers, such as CRP | 8 weeks
  Measured in mg/L
Adiponectin | 8 weeks
  Measured in μg/mL
Fibroblast growth factor 21 (FGF21). | 8 weeks
  Measured in pg/mL
Tumor necrosis factor alpha and Interleukin 6 | 8 weeks
  Measured in μg/mL
Body composition - Bioelectrical impedance | 8 weeks
  Lean mass, fat mass and adipose tissue location and distribution
Body composition - Anthropometrics | 8 weeks
  Waist, hip, neck, thigh and calf circumference measured in cm

SECONDARY OUTCOMES:
Clinical traditional and emerging markers of dietary intake | 8 weeks
  Fibroblast growth factor 21 and serum metabolites
Food cravings | 8 weeks
  Measured via self-reported questionnaire
Satiety | 8 weeks
  Assessed via serum leptin levels (ng/mL)
Cognition | 8 weeks
  Assessed via self-reported questionnaire
Impact on physical activity patterns | 8 weeks
  Assessed via accelerometry
Adherence to assigned diet | 8 weeks
  Measured via 4-day food diaries
Adherence to dietary guidelines | 8 weeks
  Measured via diet quality score assessment
Adherence to low-carbohydrate diet | 8 weeks
  Measured via blood ketones (mmol/L)
Adherence to fibre recommendations | 8 weeks
  Measured via structured questionnaires
Adherence to taking dietary supplement for low-carbohydrate, high-fat group | 8 weeks
  Measured via counting of number of multi-vitamin and mineral supplements consumed
Experience with either low-carbohydrate, high-fat or high-carbohydrate, moderate-fat diet | 8 weeks
  Assessed via semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Davies, PhD, Study Chair — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Brehm, B. et al. (2003) A randomized trial comparing a very low carbohydrate diet and a calorie-restricted low fat diet on body weight and cardiovascular risk factors in healthy women J Clin Endocrinol Metab 88(4), 1617 — http://www.ncbi.nlm.nih.gov/pubmed/12679447
- See also: Buyken, A., Goletzke, J., Joslowski, G., Felbick, A., Cheng, G., Herder, C. and Brand-Miller, J. (2014) Association between carbohydrate quality and inflammatory markers: systematic review of observational and interventional studies Am J Clin Nutr 99(4), — http://www.ncbi.nlm.nih.gov/pubmed/24552752
- See also: De Larochellière, E. et al. (2014) Visceral/epicardial adiposity in nonobese and apparently healthy young adults: association with the cardiometabolic profile Ath — http://www.ncbi.nlm.nih.gov/pubmed/24589564
- See also: Fischer, K., Pick, J., Moewes, D. and Nöthlings, U. (2015) Qualitative aspects of diet affecting visceral and subcutaneous abdominal adipose tissue: a systematic review of observational and controlled intervention studies Nutr Rev 73(4), 191-215 — http://www.ncbi.nlm.nih.gov/pubmed/26024544
- See also: Gadgil, M., Appel, L., Yeung, E., Anderson, C., Sacks, F. and Miller, E. (2013) The effects of carbohydrate, unsaturated fat, and protein intake on measures of insulin sensitivity: results from the OmniHeart trial Diabetes Care 36 (5), 1132-1137 — http://www.ncbi.nlm.nih.gov/pubmed/23223345
- See also: Gardner, C. (2012) Tailoring dietary approaches for weight loss Int J Obes Suppl 2(Suppl 1), S11-S15 — http://www.ncbi.nlm.nih.gov/pubmed/25089189
- See also: Hu, T. and Bazzano, L. (2014) The low-carbohydrate diet and cardiovascular risk factors: evidence from epidemiologic studies Nutr Metab Cardiovasc Dis 24(4), 337-343 — http://www.ncbi.nlm.nih.gov/pubmed/26393645
- See also: Hu, T., Yao, L., Reynolds, K., Niu, T., Li, S., Whelton, P., He, J., Steffen, L. and Bazzano, L. (2016) Adherence to low-carbohydrate and low-fat diets in relation to weight loss and cardiovascular risk factors Obes Sci Pract, 2(1), 24-3 — http://www.ncbi.nlm.nih.gov/pubmed/27114827
- See also: Ko, B., Park, K., Shin, S., Zaichenko, L., Davis, C., Crowell, J., Joung, H. and Mantzoros, C (2016) Diet quality and diet patterns in relation to circulating cardiometabolic biomarkers Clin Nutr. 35(2), 484-90 — http://www.ncbi.nlm.nih.gov/pubmed/25912185
- See also: Lee, M., Wu, Y. and Fried, S. (2013) Adipose tissue heterogeneity: implication of depot differences in adipose tissue for obesity complications Mol Aspects Med 34 (1), 1-11 — http://www.ncbi.nlm.nih.gov/pubmed/23068073
- See also: Lennerz, B., Alsop, D., Holsen, L., Stern, E., Rojas, R., Ebbeling, C., Goldstein, J.and Ludwig, D. (2013) Effects of dietary glycemic index on brain regions related to reward and craving in men Am J Clin Nutr 98(3), 641-647 — http://www.ncbi.nlm.nih.gov/pubmed/23803881
- See also: Allam-Ndoul, B., Guénard, F., Garneau, V., Cormier, H., Barbier, O., Pérusse, L., et al. (2016) Association between Metabolite Profiles, Metabolic Syndrome and Obesity Status. Nutrients 8(6) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4924165/
- See also: Lin, Z., Gong, Q., Wu, C., Yu, J., Lu, T., Pan, X., Lin, S. and Li, X. (2012) 'Dynamic change of serum FGF21 levels in response to glucose challenge in human J Clin Endocrinol Metab, 97(7), E1224-1228. — http://www.ncbi.nlm.nih.gov/pubmed/22539584